CLINICAL TRIAL: NCT00503425
Title: An Open Label Study to Assess the Safety and Effect on Disease Activity of MabThera in Patients With Active Rheumatoid Arthritis Who Have Had an Inadequate Response to Prior Treatment With DMARDs and/or One Anti-TNF Alpha Agent
Brief Title: A Study of MabThera (Rituximab) in Participants With Rheumatoid Arthritis Who Have Had an Inadequate Response to Disease-Modifying Antirheumatic Drugs (DMARD) and/or Anti-Tumor Necrosis Factor (Anti-TNF) Therapy.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML18606
Record Dates: First submitted 2007-07-17; First posted 2007-07-18 (Estimated); Results first posted 2016-06-23 (Estimated); Last update posted 2017-08-15 (Actual); Status verified 2017-06

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Rituximab [MabThera/Rituxan]

INTERVENTIONS:
Drug: Rituximab [MabThera/Rituxan] — 1000 mg IV on days 1 and 15

SUMMARY:
This single arm study will evaluate the safety and efficacy of MabThera in participants with active rheumatoid arthritis who have had an inadequate response to prior treatment with DMARDs and/or anti-TNF alpha agent. Participants will be treated with MabThera 1000 milligrams (mg) intravenously (IV) on days 1 and 15. Participants were followed every 8 weeks to complete 24 weeks of follow-up. After completion of the Week 24 visit, the participants were followed every 3 months for up to 18 months for an overall study duration of 24 months (104 weeks). After week 36, eligible participants who achieve moderate or good response according to the European League Against Rheumatism (EULAR) response criteria will receive re-treatment with MabThera. Participants will receive concomitant treatment with DMARDs, corticosteroids, non-steroidal anti-inflammatory drugs (NSAIDs) and analgesics throughout the study period. The anticipated time on study treatment is 2 years, and the target sample size is 200 participants.

ELIGIBILITY:
Inclusion Criteria:

During study entry

* Able and willing to give written informed consent and comply with the requirements of the study protocol;
* Participants with Rheumatoid Arthritis (RA) for at least 6 months, diagnosed according to the revised 1987 American College of Rheumatology (ACR) criteria for the classification of RA;
* Receiving treatment on an outpatient basis;
* Experienced an inadequate response to previous or current treatment with DMARDs because of toxicity or inadequate efficacy;
* Disease activity score (DAS28) greater than or equal to (>=) 3.2 at screening and baseline visit.
* Age >= 18 years;
* Participants of reproductive potential (males and females) using a reliable means of contraception (for example [e.g.] contraceptive pill, intrauterine device, physical barrier);
* Female participants with childbearing potential - a negative urine pregnancy test within two weeks prior to first rituximab treatment.

During Re-Treatment

* Achieved moderate or good response according to the EULAR response criteria during any visit including visits in the post-treatment period;
* DAS28 >=3.2;
* The participants has not been withdrawn into the safety follow-up at any time pre or post Week 24;
* 36 weeks or more have passed since the participant's first rituximab infusion;
* No evidence of any new medical condition or laboratory test results;
* In participants who were known to be positive to hepatitis B core antibody (HBcAb) - documented negative hepatitis B viral DNA (HBV-DNA) test and aspartate aminotransferase (AST)/alanine aminotransferase (ALT) less than or equal to (<=) 2.5x upper limit of normal (ULN) within the last 12 weeks;
* Female participants with childbearing potential - a negative urine pregnancy test immediately prior to treatment initiation.

Exclusion Criteria:

* Rheumatic autoimmune disease other than RA, or significant systemic involvement secondary to RA (e.g., vasculitis, pulmonary fibrosis or Felty's syndrome). Sjogren's syndrome with RA was permitted;
* Functional class IV as defined by the ACR Classification of Functional Status in RA;
* History of, or current, inflammatory joint disease other than RA (e.g., gout, reactive arthritis, psoriatic arthritis, seronegative spondyloarthropathy, Lyme disease) or other systemic rheumatic disorder disorder (e.g., inflammatory bowel disease, scleroderma, inflammatory myopathy);

Excluded Previous/Concomitant Medications

* Previous or concurrent treatment with any anti TNF-alpha therapy;
* Treatment with any investigational agent within 4 weeks of screening;
* Previous treatment with any cell depleting therapies excluding rituximab, including investigational agents;
* Immunization with a live vaccine within 4 weeks prior to the baseline visit.

Exclusions for General Safety

* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies;
* Significant cardiac or pulmonary disease (including obstructive pulmonary disease).
* Evidence of significant uncontrolled concomitant diseases such as cardiovascular disease, nervous system, pulmonary, renal, hepatic, endocrine or gastrointestinal disorders.
* Known active bacterial, viral, fungal, mycobacterial or other infection (including tuberculosis, or atypical mycobacterial disease, but excluding fungal infections of nail beds), or any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening;
* History of recurrent significant infection or history of recurrent bacterial infections;
* Primary or secondary immunodeficiency (history of, or currently active);
* Active cancer, including solid tumors and hematologic malignancies (except basal cell or squamous cell carcinoma of the skin that have been excised and cured);
* Pregnant women or nursing (breast feeding) mothers;
* Participants with lack of peripheral venous access;

Laboratory Exclusion Criteria (at Screening)

* Positive tests for hepatitis B surface antigen (HBsAg) and/or positive tests for HBcAb associated with detectable HBV-DNA or hepatitis C antibody (HCAb) and hepatitis C viral RNA (HCV-RNA).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2005-06-30 (Actual); Primary Completion 2013-05-26 (Actual); Study Completion 2013-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (16):
- Israel (16):
  - Barzilai; Rheumatology, Ashkelon
  - Assaf Harofe; Dept of Medicine B, Beer Yaakov
  - Soroka Medical Center; Reumatology, Beersheba
  - Hillel Yaffe MC; Internal C - Rheumatology, Hadera
  - Rambam Medical Center; Rheumatology, Haifa
  - Bnei Zion Medical Center; Rheumatology, Haifa
  - Carmel Hospital; Rheumatology Dept, Haifa
  - Wolfson Hospital; Rheumatology, Holon
  - Hadassah Mount Scopus Hospital; Rheumatology, Jerusalem
  - Meir Medical Center; Internal Dept A, Kfar Saba
  - Nahariya Hospital; Rheumatology Dept, Nahariya
  - Shaare Zedek Medical Center; Rheumatology Dept, Nahariya
  - EMMS Nazareth; Internal Department A, Nazareth
  - Beilinson Medical Center; Rheumatology, Petah Tikva
  - Kaplan Medical Center; Reumatology, Rehovot
  - Sourasky / Ichilov Hospital; Rheumatology, Tel Aviv

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab: Participants received rituximab (MabThera) 1000 milligrams (mg) intravenous (IV) dose on Days 1 and 15. Participants who completed the Week 36 visit and achieved moderate or good response according to the European League Against Rheumatism (EULAR) response criteria were treated again with rituximab. Rituximab was administered for up to 5 courses.
Period: Overall Study
Arm/Group | Rituximab
Started | 215
Completed | 161
Not Completed | 54
Not completed — Participant files lost | 6
Not completed — Adverse Event | 5
Not completed — Lack of Efficacy | 25
Not completed — Withdrawal by Subject | 8
Not completed — Lost to Follow-up | 3
Not completed — Death | 3
Not completed — Missing Data/Unknown | 4

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population: All participants who had received any part of infusion of study medication. Participants who prematurely withdrew from study for any reason and for whom assessment is not performed for whatever reason were also included in ITT analysis. Due to incomplete database only 209 participants were considered for analysis.
Groups:
- Rituximab: Participants received rituximab (MabThera) 1000 mg IV dose on Days 1 and 15. Participants who completed the Week 36 visit and achieved moderate or good response according to the EULAR response criteria were treated again with rituximab. Rituximab was administered for up to 5 courses.
Arm/Group | Rituximab
Number analyzed (Participants) | 209
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.6 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146
  Male | 63

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Number of participants with non-serious AEs was exclusive of SAEs.
Time Frame: Baseline up to study withdrawal or follow-up (Approximately 104 weeks)
Population: Safety population included all participants who had received any part of an infusion of study medication.
Measure: Number; unit: Participants
Arm/Group | Rituximab
Number analyzed (Participants) | 209
Participants
  AEs | 176
  SAEs | 70

2. Secondary Outcome: Mean Change From Baseline in Disease Activity Score Based on 28 Joints (DAS 28) at Week 24
Description: DAS28 score is a measure of participant's disease activity calculated using tender joint count (TJC) [28 joints], swollen joint count (SJC) [28 joints], participant's global assessment of disease activity (PGH) [visual analog scale (VAS): 0=no disease activity to 100=maximum disease activity] and erythrocyte sedimentation rate (ESR). DAS28 was calculated according to following formula: 0.56 multiplied by (*) square root (√) of TJC] plus (+) [0.28*√SJC]+[0.70*the natural logarithm (ln) ESR]+[0.014*PGH]. Total possible score of 0 to approximately 10, where higher scores represented higher disease activity. Scores below 2.6 indicated clinical remission, score of less than or equals to (</=) 3.2 indicated low disease activity, score of </=5.1 indicated moderate disease activity, scores above 5.1 indicated high or severe disease. Rituximab was administered as needed during episodes of inflammation for up to 5 courses. Change from baseline in DAS28 to Week 24 was reported for all 5 courses.
Time Frame: Baseline, Week 24
Population: ITT Population. Here, number of participants analyzed (N) signified those participants who were evaluable for this outcome and "n" signified participants with evaluable data for a specified time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rituximab
Number analyzed (Participants) | 205
Units on a scale
  Baseline (n=205) | 6.6 (1.0)
  Change at Week 24: Course 1 (n=158) | -2.3 (1.6)
  Change at Week 24: Course 2 (n=69) | -2.4 (1.3)
  Change at Week 24: Course 3 (n=30) | -2.8 (1.4)
  Change at Week 24: Course 4 (n=9) | -2.6 (1.1)
  Change at Week 24: Course 5 (n=0) | NA (NA) — Data was not analyzed as no valid data was available at week 24.
Statistical Analysis 1: Comparison: Rituximab; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Change from baseline in mean DAS28 was analyzed using paired t-test for course 1
Statistical Analysis 2: Comparison: Rituximab; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Change from baseline in mean DAS28 was analyzed using paired t-test for course 2
Statistical Analysis 3: Comparison: Rituximab; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided — Change from baseline in mean DAS28 was analyzed using paired t-test for course 3
Statistical Analysis 4: Comparison: Rituximab; Test type: Superiority or Other; p = 0.0001, t-test, 2 sided — Change from baseline in mean DAS28 was analyzed using paired t-test for course 4

3. Secondary Outcome: Percentage of Participants Whose DAS28 Improved by Greater Than (>) 1.2 at Week 24
Description: DAS28 score is a measure of participant's disease activity calculated using TJC28, SJC28, PGH [VAS: 0=no disease activity to 100=maximum disease activity] and ESR. DAS28 was calculated according to following formula: [0.56*√TJC] + [0.28*√SJC] + [0.70*ln ESR] + [0.014*PGH]. Total possible score of 0 to approximately 10, where higher scores represented higher disease activity. Scores below 2.6 indicated clinical remission, score of </= 3.2 indicated low disease activity, score of </= 5.1 indicated moderate disease activity, and scores above 5.1 indicated high or severe disease. Rituximab was administered as needed during episodes of inflammation for up to 5 courses. Change from baseline in DAS28 to Week 24 was reported for all 5 courses. Participants whose DAS28 score improved by 1.2 score were reported.
Time Frame: Week 24
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 158
Percentage of participants
  Course 1 (n=158) | 72.8
  Course 2 (n=69) | 84.1
  Course 3 (n=30) | 86.7
  Course 4 (n=9) | 77.8
  Course 5 (n=0) | NA — Data was not analyzed as no valid data was available at week 24.

4. Secondary Outcome: Percentage of Participants With EULAR DAS 28 Response at Week 24
Description: Clinical response was assessed according to EULAR categorical DAS28 response criteria, which defined clinically meaningful improvement at Week 24. EULAR response was based on change from baseline (COB) in DAS28 score and also on actual DAS28 score, at Week 24. DAS28 score= participant's disease activity calculated using TJC28, SJC28, PGH [VAS: 0=no disease activity to 100=maximum disease activity] and ESR. DAS28 was calculated by following formula: 0.56*√TJC+(0.28*√SJC)+(0.70*ln ESR)+(0.014*PGH). Total possible score=0-10, higher scores represented higher disease activity. Scores below 2.6: clinical remission, </=3.2: low disease activity, </=5.1: moderate disease activity, above 5.1: severe disease. EULAR Good response: DAS28</=3.2; COB<-1.2. Moderate response: DAS28</=3.2 or >3.2 to </=5.1 or >5.1; COB <-1.2 or <-0.6 to greater than or equal to (>/=)-1.2. No response: DAS28 </=3.2 or > 3.2 to </=5.1 or >5.1; COB <-0.6 to >/=-1.2 or >/=-0.6. EULAR response was reported for 5 courses.
Time Frame: Week 24
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Rituximab
Number analyzed (Participants) | 164
Percentage of participants
  Course 1: Good Response (n=164) | 12.8
  Course 1: Moderate Response (n=164) | 65.9
  Course 1: No Response (n=164) | 21.3
  Course 2: Good Response (n=71) | 8.5
  Course 2: Moderate Response (n=71) | 76.1
  Course 2: No Response (n=71) | 15.5
  Course 3: Good Response (n=30) | 13.3
  Course 3: Moderate Response (n=30) | 76.7
  Course 3: No Response (n=30) | 10.0
  Course 4: Good Response (n=9) | 0.0
  Course 4: Moderate Response (n=9) | 77.8
  Course 4: No Response (n=9) | 22.2
  Course 5 (n=0) | NA — Data was not analyzed as no valid data was available at week 24.

5. Secondary Outcome: Change From Baseline in Bone Density Score at Weeks 48 and 104
Description: Bone density or bone mineral density (BMD) is the amount of bone mineral in bone tissue. BMD test results are compared to the ideal or peak BMD of a healthy 30-year-old adult, and results are provided as T-score. A score of 0 means BMD is equal to the norm for a healthy young adult. Differences between observed BMD and that of the healthy young adult norm are measured in units called standard deviations (SDs). The more standard deviations below 0, indicated as negative numbers, lower the BMD higher the risk of fracture. SD + 1 to -1 indicates normal BMD; SD between -1 to -2.5 indicates low bone mass, SD -2.5 or lower indicates osteoporosis. Change in bone density was measured in participants who were not treated with biphosphonates by Dual Energy X-Ray Absorptiometry. Change in bone density was assessed at baseline and at Weeks 48 and 104. Change from baseline in bone density score was reported for all 5 courses.
Time Frame: Baseline, Weeks 48 and 104 (End of treatment)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Rituximab
Number analyzed (Participants) | 112
T-score
  Baseline: Hip T-Score (n=112) | -1.08 (1.19)
  Baseline: Spine T-Score (n=109) | -1.13 (1.26)
  Change at Week 48: Course 1, Hip T-Score ( n=14) | 0.09 (0.43)
  Change at Week 48: Course 1, Spine T-Score (n=14) | -0.03 (0.46)
  Change at Week 104: Course 1, Hip T-Score (n=11) | -0.51 (1.60)
  Change at Week 104: Course 1, Spine T-Score (n=11) | 0.45 (1.73)
  Change at Week 48: Course 2, Hip T-Score (n=0) | NA (NA) — Data was not analyzed as no valid data was available for the specified time point.
  Change at Week 48: Course 2, Spine T-Score (n=0) | NA (NA) — Data was not analyzed as no valid data was available for the specified time point.
  Change at Week 104: Course 2, Hip T-Score (n=0) | NA (NA) — Data was not analyzed as no valid data was available for the specified time point.
  Change at Week 104: Course 2, Spine T-Score (n=0) | NA (NA) — Data was not analyzed as no valid data was available for the specified time point.
  Change at Week 48: Course 3, Hip T-Score (n=0) | NA (NA) — Data was not analyzed as no valid data was available for the specified time point.
  Change at Week 48: Course 3, Spine T-Score (n=0) | NA (NA) — Data was not analyzed as no valid data was available for the specified time point.
  Change at Week 104: Course 3, Hip T-Score (n=0) | NA (NA) — Data was not analyzed as no valid data was available for the specified time point.
  Change at Week 104: Course 3, Spine T-Score (n=0) | NA (NA) — Data was not analyzed as no valid data was available for the specified time point.
  Change at Week 48: Course 4, Hip T-Score (n=0) | NA (NA) — Data was not analyzed as no valid data was available for the specified time point.
  Change at Week 48: Course 4, Spine T-Score (n=0) | NA (NA) — Data was not analyzed as no valid data was available for the specified time point.
  Change at Week 104: Course 4, Hip T-Score (n=0) | NA (NA) — Data was not analyzed as no valid data was available for the specified time point.
  Change at Week 104: Course 4, Spine T-Score (n=0) | NA (NA) — Data was not analyzed as no valid data was available for the specified time point.
  Change during Course 5 (n=0) | NA (NA) — Data was not analyzed as no valid data was available for the specified time point.

ADVERSE EVENTS:
Time Frame: Baseline up to study withdrawal or Follow-up (Approximately 104 weeks)
Description: Safety population.
Arm/Group | Rituximab
Serious Adverse Events (participants affected / at risk) | 70/209
Other Adverse Events (participants affected / at risk) | 176/209
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab (N=209)
Leukopenia (Blood and lymphatic system disorders) | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 2
Supraventricular tachycardia (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Cataract (Eye disorders) | 1
Retinal detachment (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Aphthous stomatitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Palatal disorder (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 8
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 4
Sudden death (General disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 3
Drug hypersensitivity (Immune system disorders) | 1
Abscess (Infections and infestations) | 1
Bacterial sepsis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 2
Otitis externa (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 4
Pulmonary tuberculosis (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Femur fracture (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 2
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2
Periprosthetic fracture (Injury, poisoning and procedural complications) | 2
Road traffic accident (Injury, poisoning and procedural complications) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 2
Toxicity to various agents (Injury, poisoning and procedural complications) | 1
Endoscopy (Investigations) | 1
Endoscopy upper gastrointestinal tract (Investigations) | 1
Fibrin D dimer (Investigations) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 11
Aphasia (Nervous system disorders) | 1
Cerebrovascular disorder (Nervous system disorders) | 2
Hemiparesis (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Radicular pain (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 4
Abortion (Pregnancy, puerperium and perinatal conditions) | 1
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 4
Anxiety (Psychiatric disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Joint manipulation (Surgical and medical procedures) | 1
Pain management (Surgical and medical procedures) | 1
Polypectomy (Surgical and medical procedures) | 1
Spinal laminectomy (Surgical and medical procedures) | 1
Deep vein thrombosis (Vascular disorders) | 1
Raynaud's phenomenon (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab (N=209)
Anaemia (Blood and lymphatic system disorders) | 11
Chest pain (General disorders) | 14
Pyrexia (General disorders) | 12
Upper respiratory tract infection (Infections and infestations) | 21
Urinary tract infection (Infections and infestations) | 15
Hyperlipidaemia (Metabolism and nutrition disorders) | 12
Vitamin D deficiency (Metabolism and nutrition disorders) | 22
Arthralgia (Musculoskeletal and connective tissue disorders) | 12
Back pain (Musculoskeletal and connective tissue disorders) | 28
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 25
Headache (Nervous system disorders) | 20
Rash (Skin and subcutaneous tissue disorders) | 14
Hypertension (Vascular disorders) | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.